CLINICAL TRIAL: NCT02982655
Title: A Multi-center Randomised Controlled Trial to Explore the Ideal Individualized Anti-hypertension Strategies in Patients With Severe Stroke at Acute Stage
Brief Title: Controlling Hypertension After Severe Cerebrovascular Event
Acronym: CHASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Tang-Du Hospital (Other); Xi'an Central Hospital (Other); Shaanxi Provincial People's Hospital (Other); Hanzhong Central Hospital (Other); Yan'an University Affiliated Hospital (Other); Xiangyang Central Hospital (Other); Xi'an 141 Hospital (Unknown); Shangluo Central Hospital (Other); 215 Hospital of Shaanxi NI (Other); Yulin No.2 Hospital (Other); Yulin No.1 Hospital (Unknown); Ankang Central Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xi'an Gaoxin Hospital (Other); 521 Hospital of NORINCO Group (Other); Xi'an No.3 Hospital (Other Government); Xi'an No.4 Hospital (Unknown); Xi'an No.9 Hospital (Unknown); Xi'an XD Group Hospital (Unknown); Xi'an Traditional Chinese Medicine Hospital (Other); Baoji Central Hospital (Other); Weinan Central Hospital (Other); Tongchuan Mining Hospital (Unknown); Tongchuan People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20162085-2
Record Dates: First submitted 2016-11-27; First posted 2016-12-05 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2018-09

CONDITIONS: Severe Stroke; Acute Stroke; Hypertension
Keywords: Severe Stroke; Acute Stroke; Antihypertension; mortality; disability; clinical trial
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized BP lowering (Experimental): Management policy is to lower the systolic or diastolic BP by 10-15% within 2 hours of randomization and sustained for 7 days. Sites were provided with protocols for different intravenous agents and used whichever routinely available drugs were in their hospital.
  Interventions: Procedure: Individualized BP lowering
- Guideline recommended BP lowering (Active Comparator): Patients received management of BP based on the standard guidelines at the time, as published by the Chinese Society of Neurology (CSN) in 2014. The attending clinician may consider commencing BP treatment and sustained for 7 days if the systolic BP > 200 mmHg or diastolic BP >110 mmHg in patients with ischemic stroke, and systolic BP > 180 mmHg or diastolic BP > 110 mmHg in patients with cerebral hemorrhage.
  Interventions: Procedure: Individualized BP lowering

INTERVENTIONS:
Procedure: Individualized BP lowering

SUMMARY:
The purpose of this academic lead study is to explore ideal blood pressure targets and optimum individualized anti-hypertension strategies in acute severe stroke.

DETAILED DESCRIPTION:
Of high mortality and morbidity, severe stroke is associated with devastating damages in neurologic, respiratory, circulatory and many other systems. The outcomes of patients with severe stroke depend largely on medical strategies on acute stage, especially on blood pressure (BP) management. Unfortunately, so far no ideal BP range has been scientifically determined for patients with acute severe stroke.

The CHASE study aims to provide reliable data on the effects of individualized anti-hypertension strategy in patients with acute severe stroke (target recruitment 250) compared to standard guideline-based management of BP (target recruitment 250). Patients presenting with acute (<72h) severe stroke (GCS ≦ 12 or NIHSS ≧ 11) and elevated BP (systolic blood pressure ≧150 mmHg or diastolic blood pressure ≧ 100 mmHg) will be randomly assigned to individualized anti-hypertension treatment or guideline-based treatment for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. the randomly assigned BP-lowering regimen is able to be commenced within 72 h after the onset of stroke (ischemic or hemorrhagic), confirmed by a computed tomography (CT) or magnetic resonance imaging (MRI) scan of the brain (if the precise timing of the onset of symptoms or signs of the qualifying event is unknown, then the time of onset will be taken as the last time the patient was known to be well);
3. GCS on admission ≤ 12 or NIHSS on admission ≥ 11;
4. there are at least two SBP measurements of ≥ 150 and ≤ 210 mmHg, recorded ≥5 min apart (patients with an initial SBP < 150 mmHg may be randomized when the SBP fulfils entry criteria on rechecking up to 72 h after the onset of stroke);
5. written informed consent is able to be obtained directly from the patient or an appropriate surrogate, based on local ethics committee recommendations.

Exclusion Criteria:

1. patients who have received thrombolytic therapy, embolectomy, or decompressive craniectomy for the current stroke;
2. patients with subarachnoid hemorrhage;
3. known definite contraindication to acute BP lowering (e.g. known severe carotid, vertebral, or cerebral arterial stenosis, Moyamoya disease or Takayasu's arteritis, high grade stenotic valvular heart disease);
4. secondary to a structural abnormality in the brain (e.g. an arteriovenous malformation, intracranial aneurysm, tumor, or trauma);
5. unstable vital signs and requiring the use of vasoactive agents;
6. known existing dementia or prestroke disability (e.g. score 3-5 on the modified Rankin scale);
7. concomitant medical illness that would interfere with the outcome assessments and/or follow-up (advanced cancer; severe pulmonary dysfunction [forced expiratory volume in 1 s < 50%]; severe cardiac dysfunction [ejection fraction ≤ 50%]; severe hepatic failure [Child-Pugh score ≥ 7]; severe renal failure [glomerular filtration rate ≤ 30 mL/min or serum creatinine ≥ 4 mg/dL]);
8. patients who are currently participating in other investigational trials;
9. patients who are considered to have a high likelihood of not adhering to the study treatment or the follow-up regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Death or major disability (the modified Rankin scale ≥ 3) | 3 months after onset
  Components of modified Rankin Scale score:0,No symptoms;1,No significant disability despite symptoms;2,Slight disability;3,Moderate disability requiring some help, but able to walk without assistance;4,Moderate severe disability;5,Severe disability;6,Death.

SECONDARY OUTCOMES:
Ability of activities of daily living at day 90 of enrollment (defined by Barthel Index) | 3 months after onset
  Barthel Index is a 100-point scale (0-100), where higher scores indicate better ability of activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, PhD, Study Director — Department of Neurology, Xijing Hospital, Fourth Military Medical University
Locations (26):
- China (26):
  - Ankang Central Hospital, Ankang, Shaanxi
  - Baoji Central Hospital, Baoji, Shaanxi
  - Hanzhong Central Hospital, Hanzhong, Shaanxi
  - Shangluo Central Hospital, Shangluo, Shaanxi
  - Tongchuan Mining Hospital, Tongchuan, Shaanxi
  - Tongchuan People's Hospital, Tongchuan, Shaanxi
  - Weinan Central Hospital, Weinan, Shaanxi
  - Xi'an 141 Hospital, Xi'an, Shaanxi
  - Department of Neurology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - 521 Hospital of NORINCO Group, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Xi'an Gaoxin Hospital, Xi'an, Shaanxi
  - Xi'an No.3 Hospital, Xi'an, Shaanxi
  - Xi'an No.4 Hospital, Xi'an, Shaanxi
  - Xi'an No.9 Hospital, Xi'an, Shaanxi
  - Xi'an Traditional Chinese Medicine Hospital, Xi'an, Shaanxi
  - Xi'an XD Group Hospital, Xi'an, Shaanxi
  - Xianyang Central Hospital, Xianyang, Shaanxi
  - 215 Hospital of Shaanxi NI, Xianyang, Shaanxi
  - Yan'an University Affiliated Hospital, Ya'an, Shaanxi
  - Yulin No.2 Hospital, Yulin, Shaanxi
  - Yulin No.1 Hospital, Yulin, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sandset EC, Bath PM, Boysen G, Jatuzis D, Korv J, Luders S, Murray GD, Richter PS, Roine RO, Terent A, Thijs V, Berge E; SCAST Study Group. The angiotensin-receptor blocker candesartan for treatment of acute stroke (SCAST): a randomised, placebo-controlled, double-blind trial. Lancet. 2011 Feb 26;377(9767):741-50. doi: 10.1016/S0140-6736(11)60104-9. PMID 21316752
- [Background] Vemmos KN, Spengos K, Tsivgoulis G, Zakopoulos N, Manios E, Kotsis V, Daffertshofer M, Vassilopoulos D. Factors influencing acute blood pressure values in stroke subtypes. J Hum Hypertens. 2004 Apr;18(4):253-9. doi: 10.1038/sj.jhh.1001662. PMID 15037874
- [Background] AlSibai A, Qureshi AI. Management of Acute Hypertensive Response in Patients With Ischemic Stroke. Neurohospitalist. 2016 Jul;6(3):122-9. doi: 10.1177/1941874416630029. Epub 2016 Apr 21. PMID 27366297
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Result] CAST: randomised placebo-controlled trial of early aspirin use in 20,000 patients with acute ischaemic stroke. CAST (Chinese Acute Stroke Trial) Collaborative Group. Lancet. 1997 Jun 7;349(9066):1641-9. PMID 9186381
- [Result] Qureshi AI, Ezzeddine MA, Nasar A, Suri MF, Kirmani JF, Hussein HM, Divani AA, Reddi AS. Prevalence of elevated blood pressure in 563,704 adult patients with stroke presenting to the ED in the United States. Am J Emerg Med. 2007 Jan;25(1):32-8. doi: 10.1016/j.ajem.2006.07.008. PMID 17157679
- [Result] Castillo J, Leira R, Garcia MM, Serena J, Blanco M, Davalos A. Blood pressure decrease during the acute phase of ischemic stroke is associated with brain injury and poor stroke outcome. Stroke. 2004 Feb;35(2):520-6. doi: 10.1161/01.STR.0000109769.22917.B0. Epub 2004 Jan 15. PMID 14726553
- [Result] Schrader J, Luders S, Kulschewski A, Berger J, Zidek W, Treib J, Einhaupl K, Diener HC, Dominiak P; Acute Candesartan Cilexetil Therapy in Stroke Survivors Study Group. The ACCESS Study: evaluation of Acute Candesartan Cilexetil Therapy in Stroke Survivors. Stroke. 2003 Jul;34(7):1699-703. doi: 10.1161/01.STR.0000075777.18006.89. Epub 2003 Jun 19. PMID 12817109
- [Result] Potter JF, Robinson TG, Ford GA, Mistri A, James M, Chernova J, Jagger C. Controlling hypertension and hypotension immediately post-stroke (CHHIPS): a randomised, placebo-controlled, double-blind pilot trial. Lancet Neurol. 2009 Jan;8(1):48-56. doi: 10.1016/S1474-4422(08)70263-1. Epub 2008 Dec 4. PMID 19058760
- [Result] Robinson TG, Potter JF, Ford GA, Bulpitt CJ, Chernova J, Jagger C, James MA, Knight J, Markus HS, Mistri AK, Poulter NR; COSSACS Investigators. Effects of antihypertensive treatment after acute stroke in the Continue or Stop Post-Stroke Antihypertensives Collaborative Study (COSSACS): a prospective, randomised, open, blinded-endpoint trial. Lancet Neurol. 2010 Aug;9(8):767-75. doi: 10.1016/S1474-4422(10)70163-0. PMID 20621562
- [Result] He J, Zhang Y, Xu T, Zhao Q, Wang D, Chen CS, Tong W, Liu C, Xu T, Ju Z, Peng Y, Peng H, Li Q, Geng D, Zhang J, Li D, Zhang F, Guo L, Sun Y, Wang X, Cui Y, Li Y, Ma D, Yang G, Gao Y, Yuan X, Bazzano LA, Chen J; CATIS Investigators. Effects of immediate blood pressure reduction on death and major disability in patients with acute ischemic stroke: the CATIS randomized clinical trial. JAMA. 2014 Feb 5;311(5):479-89. doi: 10.1001/jama.2013.282543. PMID 24240777
- [Result] Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J; INTERACT Investigators. Intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT): a randomised pilot trial. Lancet Neurol. 2008 May;7(5):391-9. doi: 10.1016/S1474-4422(08)70069-3. Epub 2008 Apr 7. PMID 18396107
- [Result] Anderson CS, Heeley E, Huang Y, Wang J, Stapf C, Delcourt C, Lindley R, Robinson T, Lavados P, Neal B, Hata J, Arima H, Parsons M, Li Y, Wang J, Heritier S, Li Q, Woodward M, Simes RJ, Davis SM, Chalmers J; INTERACT2 Investigators. Rapid blood-pressure lowering in patients with acute intracerebral hemorrhage. N Engl J Med. 2013 Jun 20;368(25):2355-65. doi: 10.1056/NEJMoa1214609. Epub 2013 May 29. PMID 23713578
- [Derived] Yuan F, Yang F, Zhao J, Fu F, Liu Y, Xue C, Wang K, Yuan X, Li D, Liu Q, Zhang W, Jia Y, He J, Zhou J, Wang X, Lv H, Huo K, Li Z, Zhang B, Wang C, Li L, Li H, Jiang W. Controlling Hypertension After Severe Cerebrovascular Event (CHASE): A randomized, multicenter, controlled study. Int J Stroke. 2021 Jun;16(4):456-465. doi: 10.1177/1747493020932784. Epub 2020 Jun 11. PMID 32525464
- [Derived] Yuan F, Yang F, Xue C, Wang K, Liu Q, Zhou J, Fu F, Wang X, Zhang W, Liu Y, Huo K, Lv H, Jiang W; CHASE Study Group. Controlling Hypertension After Severe Cerebrovascular Event (CHASE): study protocol for a randomized controlled trial. Trials. 2018 Feb 21;19(1):130. doi: 10.1186/s13063-018-2530-x. PMID 29467025